CLINICAL TRIAL: NCT04310878
Title: Gaps Between Evidence and Practice in Prevention of Surgical Site Infection in Spain: A Survey of the Observatory of Infection in Surgery
Brief Title: Gaps Between Evidence and Practice in Prevention of Surgical Site Infection in Spain
Acronym: SurveyOIC
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Other Study IDs: OIC Survey3
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-03

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Preventative measures
MeSH Terms: conditions — Surgical Wound Infection | interventions — Surgeons

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey among perioperative nurses and surgeons — Online survey

SUMMARY:
Web-based survey to members of 10 Spanish Associations of surgical nurses and surgeons of different specialities to know the application of preventative measures for surgical site infection.

DETAILED DESCRIPTION:
A web-based survey to the members of the Colorectal Chapter of 10 Spanish Associations of surgical nurses and surgeons of different specialities. A link to the web page containing the survey will be disseminated via email, newsletter and Twitter.

A board from the Surgical Infection Section did a review of evidence and previous guidelines to be used in the evaluation of the results. The most recent clinical practice guidelines have been analysed. According to the review, the preventive measures analysed in the survey have been distributed into two groups: high or low level of evidence.

The survey aim to assess knowledge, beliefs, and practices of attending nurses and surgeons on preventative measures. Furthermore, the questions address the level of accordance between their beliefs and the protocols or the usual practice of their units. The agreement rate between the beliefs and usual practice of all respondents will be calculated on a scale from 0 to 100. For discussion, the responses on the implementation of major surgical site infection (SSI) prevention measures will be compared with the recommendations of the expert group.

The results will be expressed in percentages on the total answers obtained. Responses will be entered into a computerized database that will be analysed using an specific program. The results will be analysed using the chi-square test with statistical significance defined as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Nurses and surgeons pertaining to invited societies

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Perioperative nurses and surgeons of 11 invited Spanish societies
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Awareness of practice | 2020
  Percentage of responders who use each preventive measures for surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Josep Badia-Perez, MD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No